CLINICAL TRIAL: NCT04357457
Title: Efficacy of Intravenous Almitrine in Reducing the Need for Mechanical Ventilation in Patients With Hypoxemic Acute Respiratory Failure Due to Covid-19-related Pneumonia: a Randomized Controlled Double-blind Study From the Skip-icu Consortium
Brief Title: Efficacy of Intravenous Almitrine in Reducing the Need for Mechanical Ventilation in Patients With Hypoxemic Acute Respiratory Failure Due to Covid-19-related Pneumonia
Acronym: AIRVM-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200461; 2020-001909-22 (EudraCT Number)
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Covid 19; Hypoxemic Respiratory Failure
Keywords: Almitrine; HYPOXEMIC ACUTE RESPIRATORY FAILURE; COVID-19; COVID-19 pneumonia
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Almitrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almitrine (Experimental)
  Interventions: Drug: Almitrine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Almitrine — Intravenous almitrine at a dose of 2 µg.kg-1.min-1 during 5 days
  Arms: Almitrine
Drug: Placebo — Intravenous glucose 5% during 5 days
  Arms: Placebo

SUMMARY:
The COVID-19 outbreak is associated with a surge in ICU bed requirement and substantial mortality (estimated between 0.5% and 1%). Admission in the intensive care unit (ICU) and need for mechanical ventilation is reportedly associated with an estimated hospital mortality of more than 30%. Furthermore, the surge in ICU bed requirement is a worldwide-shared issue, leading to sub-optimal ICU management.

In acute respiratory failure due to COVID-19-related pneumonia, vasoplegia with vascular enlargement inside the lung lesions and dilation of small vessels seen on chest CT scan largely account for severe hypoxemia whose physiological response is hyperventilation leading to hypocapnia. Almitrine, initially described to reduce intrapulmonary shunt by enhancement of hypoxic pulmonary vasoconstriction in combination with inhaled nitric oxide (iNO), redistributes pulmonary blood flow from shunt areas to lung units with normal ventilation/perfusion (VA/Q) ratio. Low dose of intravenous almitrine (2 µg.kg-1.min-1) alone also improves oxygenation (without combination with iNO) by selective pulmonary vasoconstriction of precapillary pulmonary arteries perfusing lung areas exposed to a hypoxic challenge with a slight increase in mean arterial pulmonary. Therefore, our hypothesis is that 5 days of low dose of almitrine therapy may improve the ventilation-perfusion (VA/Q) ratio at a relatively early stage of this specific lung disease and limit respiratory worsening and subsequent need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged 80 years or less
* COVID-19 diagnosis defined as either positive RT-PCR for SARS-CoV-2 or COVID-19 compatible or typical chest CT pattern or positive serology for COVID-19 antibodies
* Hypoxemic acute respiratory failure with the following criteria: oxygen saturation level of 92% or less, as measured by pulsed oximetry (SpO2) under oxygen therapy with an oxygen rate of 6L/min or more.
* Hospital admission for COVID-19 within 14 days
* Patients affiliated

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Pregnancy or breastfeeding woman
* Known Hepatic failure (PT <50%, Factor V < 50%)
* Last known Plasma total bilirubin > 21 μmol/L
* Lactate level > 4 mmol/L
* ALT and AST levels greater than 3 times the upper limit
* Pulmonary hypertension (PAPs ≥37 mmHG and/or VmaxIT ≥ 2,9 m/s) or right ventricular dysfunction
* History of pulmonary embolism
* Diagnosis of pulmonary embolism during the current hospitalization or on-going anticoagulant therapy at curative dose for thromboembolism when hospitalized
* PaCO2 > 45 mmHg
* Exacerbation of asthma or chronic respiratory failure
* Cardiogenic pulmonary oedema
* Systolic blood pressure of 90 mmHg or less, or use of vasopressors
* Urgent need for endotracheal intubation at the discretion of the treating physician
* Do-not-intubate order or estimated life expectancy less than 6 months
* Participation in another interventional research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Rate of endotracheal intubation | 7 days
  Endotracheal intubation within 7 days after randomization Death will be considered as a failure (endotracheal intubation).

SECONDARY OUTCOMES:
28-day mortality | 28 days
In-hospital mortality | 28-day
Number of ventilator-free days | 28 days
Number of days in the ICU | 28 days
Number of days in the hospital | 28 days
Discontinuation rate of the treatment | 28 days
  safety assessment: discontinuation rate of the treatment for arterial lactate more than 4 mmol/L, ALT/AST levels greater than 3 times the upper limit, and diagnosis of pulmonary arterial hypertension or acute cor pulmonale documented by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Yes, upon request, after approval by the primary investigator and clinical research platform of East Paris. For the purpose of IPD meta-analysis, or secondary analysis. Unidentifying data will be shared.

REFERENCES:
- [Derived] Kalfon P, Payen JF, Rousseau A, Chousterman B, Cachanado M, Tibi A, Audibert J, Depret F, Constantin JM, Weiss E, Remerand F, Freund Y, Simon T, Riou B. Effect of intravenous almitrine on intubation or mortality in patients with COVID-19 acute hypoxemic respiratory failure: A multicentre, randomised, double-blind, placebo-controlled trial. EClinicalMedicine. 2022 Oct;52:101663. doi: 10.1016/j.eclinm.2022.101663. Epub 2022 Sep 21. PMID 36157895